CLINICAL TRIAL: NCT05764434
Title: Spinal Cord Gray and White Matter Imaging in Amyotrophic Lateral Sclerosis
Brief Title: ALS Spinal Cord Gray and White Matter Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Regina Schlaeger, PD Dr., University Hospital, Basel, Switzerland
Other Study IDs: ALS_SC_MRI
Record Dates: First submitted 2023-02-27; First posted 2023-03-10 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Spinal Cord Magnetic Resonance Imaging
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Amyotrophic Lateral Sclerosis: Patients with a possible, probable, or definite diagnosis of Amyotrophic Lateral Sclerosis according to the El Escorial Criteria.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging
- Healthy Control Persons: Healthy control persons matching the ALS patient group in sex and age
  Interventions: Diagnostic Test: Magnetic Resonance Imaging
- Patients with other Motor Neuron Diseases: Patients with Motor Neuron Diseases other than ALS
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Magnetic Resonance Imaging of the spinal cord using radially acquired Averaged Magnetization Inversion Recovery Acquisitions (rAMIRA)

SUMMARY:
This study aims to measure in vivo the spinal cord gray and white matter in patients with Amyotrophic Lateral Sclerosis and healthy persons that match the patients' age and sex using rAMIRA imaging, a novel Magnetic Resonance Imaging (MRI) method. Patients and healthy control persons prospectively undergo MRI examinations, clinical examinations including assessments of disability, and tests of muscle force using hand held dynamometry. Serum markers of neuro-axonal injury are also assessed.

Examinations for patients and healthy control persons are scheduled every six months over a time span of two years.

ELIGIBILITY:
Inclusion Criteria (patients):

1. 18 years or older
2. neurologist-confirmed possible, probable or definite ALS acc. to El Escorial criteria
3. at baseline: able to lie in an MRI scanner for one hour

Exclusion Criteria (patients):

1. active other neurological or neuromuscular condition explaining the symptoms or a significant part of it
2. other neurological or neuromuscular conditions interfering with the examinations
3. severe cervical spinal stenosis or other relevant disease of the spine or spinal cord that may interfere with study procedures or that may impact the cord segments imaged in this study
4. other severe chronic disease
5. pregnancy
6. general contraindications against MRI scanning (e.g. metal implants, pacemakers)
7. not able to read the patient information due to language barriers (patient information in English and French may be provided)
8. major cognitive deficit impacting the ability to read and understand the patient information and/or to follow the instructions of the study personnel

Inclusion criteria (healthy control persons):

1. 18 years or older
2. able to lie in MRI scanner for one hour

Exclusion criteria (healthy control persons):

1. neurological or neuromuscular conditions
2. other severe chronic disease
3. pregnancy
4. general contraindications against MRI scanning (e.g. metal implants, pacemakers)
5. relevant cervical spinal canal stenosis or other relevant disease of the spine or spinal cord that may interfere with study procedures or that may impact the cord segments imaged in this study
6. not able to read the patient information due to language barriers (patient information in English and French may be provided)

Inclusion criteria (patients with Motor Neuron Diseases other than ALS):

1. 18 years or older
2. neurologist-confirmed Motor Neuron Disease (not ALS)
3. able to lie in MRI scanner for one hour

Exclusion criteria (patients with Motor Neuron Diseases other than ALS):

1. other severe neurologic disease
2. other severe chronic disease
3. pregnancy
4. general contraindications against MRI scanning (e.g. metal implants, pacemakers)
5. relevant cervical spinal canal stenosis or other relevant disease of the spine or spinal cord that may interfere with study procedures or that may impact the cord segments imaged in this study
6. not able to read the patient information due to language barriers (patient information in English and French may be provided)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with possible, probable, and definite Amyotrophic Lateral Sclerosis acc. to the El Escorial aged 18 years or older can participate in this study. Healthy control persons are chosen to individually match the included patients. Additionally, patients with other motor neuron diseases (not ALS) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Spinal Cord Gray Matter Baseline | baseline
  Spinal cord gray matter cross-sectional area in mm2
Spinal Cord Gray Matter 6 month follow-up | 6 month follow-up
  Spinal cord gray matter cross-sectional area in mm2
Spinal Cord Gray Matter 12 month follow-up | 12 month follow-up
  Spinal cord gray matter cross-sectional area in mm2
Spinal Cord Gray Matter 18 month follow-up | 18 month follow-up
  Spinal cord gray matter cross-sectional area in mm2
Spinal Cord Gray Matter 24 month follow-up | 24 month follow-up
  Spinal cord gray matter cross-sectional area in mm2

SECONDARY OUTCOMES:
Spinal Cord White Matter | baseline, months 6, 12, 18 and 24
  Spinal cord white matter cross-sectional area in mm2
Spinal Cord Total Area | baseline, months 6, 12, 18 and 24
  Total spinal cord cross-sectional area in mm2
ALS Functional Rating Scale | baseline, months 6, 12, 18 and 24
  ALS Functional Rating Scale (ALSFRS-R)
Neurofilament Light Chain Levels | baseline, months 6, 12, 18 and 24
  Neurofilament Light Chain Levels (pg/ml)
Sniff nasal inspiratory pressure | baseline, months 6, 12, 18 and 24
  Sniff nasal inspiratory pressure (SNIP) (cmH2O)
Segmental Muscle Force | baseline, months 6, 12, 18 and 24
  Segmental Muscle Force assessed by hand-held dynamometry (N)
MUNIX | baseline, months 6, 12, 18 and 24
  Motor Unit Number Index (MUNIX) in selected muscles

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No